CLINICAL TRIAL: NCT05190627
Title: Phase II Clinical Trial Evaluating the Effect of Loratadine Associated to Rapamicyn in Patients With Lymphangioleiomyomatosis
Brief Title: Effect of Loratadine in Lymphangioleiomyomatosis
Acronym: LORALAM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut d'Investigació Biomèdica de Bellvitge (Other)
Responsible Party: Principal Investigator, Maria Molina, Chief of Interstitial Lung Diseases Unit, Respiratory Department. Associated Professor (University of Barcelona), Institut d'Investigació Biomèdica de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LORALAM
Record Dates: First submitted 2021-12-11; First posted 2022-01-13 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Lymphangioleiomyomatosis
Keywords: LAM; Rapamycin; Loratadine
MeSH Terms: conditions — Lymphangioleiomyomatosis | interventions — Loratadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Loratadine treatment on rapamycin (Experimental): Loratadine (oral administration, daily dose 10mg) in LAM patients that are treated with rapamycin
  Interventions: Drug: Loratadine
- Placebo treatment on rapamycin (Placebo Comparator): Placebo (oral administration, daily dose 10 mg) in LAM patients that are treated with rapamycin
  Interventions: Drug: Placebo 10mg/day added to rapamycin for 12 months

INTERVENTIONS:
Drug: Loratadine — Loratadine 10mg/day added to rapamycin for 12 months
  Other Names: Clarytine
  Arms: Loratadine treatment on rapamycin
Drug: Placebo 10mg/day added to rapamycin for 12 months — Placebo in the same type of capsule than the experimental drug
  Arms: Placebo treatment on rapamycin

SUMMARY:
INTRODUCTION: LAM is a rare and lethal disease characterized by progressive cystic lung destruction. Inhibition of mTOR with rapamycin is the current standard of care (SOC), which can slow-down disease. Plasma major histamine metabolite (Methylimidazoleacetic acid [MIAA]) is increased in LAM. Loratadine is a histamine receptor antagonist (HR1), which inhibits LAM cell proliferation. Therefore, a novel phase-II clinical trial for assessing safety and potential benefits of loratadine in LAM has been initiated.

METHODS: LORALAM clinical trial, phase-II, double-blind, randomized, placebo controlled, parallel-group, multicentre study initiates recruitment in July 2020. Enrollment plan includes 62 subjects with LAM on treatment with rapamycin ≥3 months, randomized 1:1 to add oral loratadine 10mg/day or placebo, once daily, for 52 weeks. Recruitment will end in June 2021. The primary endpoints are 1) to assess the safety profile of loratadine associated with rapamycin, 2) lung function decline after 52 weeks of treatment. The secondary endpoints are a) quality of life and progression free-survival time, b) changes in the established LAM serum biomarker VEGFD, c) the utility of MIAA for monitoring disease progression and biological treatment effect.

ETHICS AND DISSEMINATION: The study will be carried out in accordance with Good Clinical Practice guidelines, Declaration of Helsinki principles, and each ethical committee. This clinical trial contemplates the possibility of increasing the number of centers and including patients from patient support groups (LAM foundation, AELAM)

DETAILED DESCRIPTION:
Lymphangioleiomyomatosis (LAM) is a rare and lethal lung disease affecting almost exclusively women of childbearing age and characterized by progressive cystic lung destruction. LAM results from germline and somatic loss-of-function mutations in the tuberous sclerosis complex 1 and 2 genes (TSC1/2), and therefore diseased cells show abnormal activation of the mechanistic target of rapamycin (mTOR). Inhibition of mTOR with rapamycin (also known as sirolimus) is the current standard of care. However, this therapy does not fully kill LAM cells, shows variable tolerability and treatment answer. Therefore, sirolimus has slowed-down disease progression but young patients still need lung transplantation despite treatment. In addition, LAM diagnosis and clinical monitoring is also challenging due to the heterogeneity of symptoms and insufficiency of non-invasive tests. Here, guided by comprehensive preclinical data obtained in the context of a Spanish research network for LAM, and with the support of the national Association of LAM patients (AELAM), the investigators propose a phase-II clinical trial for assessing if the tricyclic antihistamine loratadine is effective in slowing the progression of lung disease in LAM. Loratadine is an histamine receptor 1 (HR1) antagonist, widely used for allergic process, that also acts through different intracellular signaling, including Akt/MITF and PKCBII-tyrosine kinase. Recent studies have demonstrated that co-treatment with loratadine sensitize KBV20C resistant cells to vincristine, which improve the onco-therapeutical effect. The primary study objective is to assess the safety profile of loratadine 10 mg/day associated with the current standard treatment (sirolimus) and its potential benefit abrogating the lung function decline after 52 weeks of treatment. The secondary objectives include; a) an assessment of quality of life and progression free-survival time, and, b) to determine the clinical usefulness of the major histamine-derived metabolite methylimidazoleacetic acid (MIAA) for monitoring of disease progression and biological treatment effect.

ELIGIBILITY:
Inclusion Criteria:

* 1. Written informed consent consistent with GCP and local laws signed prior to entry into the study.

  2. Patients with LAM and > 18 years-old with:
* FEV1 > 35% and DLCO > 20%
* Oxygen saturation (SpO2) > 85% by pulse oximetry while breathing ambient air at rest
* Patients with a definite diagnosis consistent with LAM prior to screening based on International consensus criteria within 10 years prior to randomization
* HRCT within 12 months prior to randomization with central reading demonstrating a radiological pattern suggesting LAM and some other criteria for initiating sirolimus (symptoms, FEV1 decline or the presence of abdominal lynphangioleiomiomas).

Exclusion Criteria:

* Concomitant use of other HR1 antagonist
* Hypersensitivity to HR1 antagonists
* Current smoker or ex-smoker having quit smoking < 4 months prior to firs screening visit - Use of systemic immunosuppressants or chemotherapy within 30 days of screening.
* Receiving oral corticosteroids>15mg/day, vasodilator therapies for pulmonary hypertension (e.g., bosentan), unapproved and/or investigational therapies for LAM or administration of such therapies within 4 weeks of initial screening.
* At baseline/screening visit, values of liver transaminases above 3 times upper limit, alkaline phosphatase above 2.5 times upper limit, or bilirubin above 1.5 times upper limit
* Creatinine clearance (CrCl)<60ml/min (determined by Cockcroft-Gault Equation) at baseline/ screening visit.
* Patients treated with strong inhibitors and inducers of CYP either during the study or 14 days prior to enrolment in the study: antifungals (e.g., ketoconazole, itraconazole), clarithromycin, telithromycin, cobicistat, protease inhibitors (e.g., atazanavir, ritonavir, and saquinavir) and grapefruit juice, phenytoin, carbamazepine, barbiturates, rifampin.
* Current allergic asthma or other major allergic diseases that requires different daily anti- histaminic treatment.
* History of coexistent and clinically significant (in the opinion of the Investigator) chronic obstructive pulmonary disease (COPD), bronchiectasis, asthma, inadequately treated sleep- disordered breathing, or any clinically significant pulmonary diseases other than LAM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (safety) of loratadine in combination with sirolimus after 52 weeks of treatment | 52 weeks
  To compare the incidence of adverse events in LAM patients treated with sirolimus and loratadine versus sirolimus alone. Any adverse event related to both drugs, including nausea, diarrhea, stomach discomfort, vomiting, headache and liver hipertransaminasemia, will be evaluated.

SECONDARY OUTCOMES:
To evaluate the effect of loratadine associated with sirolimus on quality of life measured by the Saint George's Questionnaire | 52 weeks
  The Saint George's Questionnaire is one of the most validated questionnaires in respiratory diseases that evaluates three dimensions; symptoms, activity and disease impact, and the total score ranges from 0 (worse situation) to 100 (best situation).
Study-drug discontinuation | 52 weeks
  To compare the rate of study-drug discontinuation during the study in both arms
Serum levels of sirolimus | 52 weeks
  Analyzing the number of patients that maintain the serum levels of sirolimus on window range that is considered therapeutic and safe (5-15 pg).
To evaluate the effect of loratadine associated with sirolimus on progression-free survival time | 52 weeks
  Progression-free survival time, which will be considered when some of these events are present: FEV1 decrease > 10%, DLCO decrease > 15%, lung transplant, death.
To evaluate the effect of loratadine associated with sirolimus on hospitalization rate | 52 weeks
  Hospitalization. Registration of any cause of hospitalization.
To evaluate the effect of loratadine associated with sirolimus on serum biomarkers | 52 weeks
  Serum biomarkers: measuring changes on the single established biomarker to date (VEGF-D)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Molina-Molina, MD, PhD, Study Director — Institut d'Investigació Biomèdica de Bellvitge
Locations (6):
- Spain (6):
  - University Hospital of Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital La Princes, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Marqués de Valdecillas, Santander
  - Hospital Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: IDIBELL webpage — http://idibell.cat